CLINICAL TRIAL: NCT06646250
Title: NeoDoppler: New Ultrasound Technology for Continuous Monitoring of Cerebral Blood Flow in Infants
Brief Title: NeoDoppler: New Ultrasound Technology for Continuous Monitoring of Cerebral Circulation Pilot
Acronym: CE-NeoDoppler
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/314
Record Dates: First submitted 2024-08-23; First posted 2024-10-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Preterm; Patent Ductus Arteriosus; Sepsis; Asphyxia; Stroke; Pulmonary Hypertension; Congenital Heart Disease
Keywords: Cerebral Doppler; Monitoring; Continuous; Neonate
MeSH Terms: conditions — Premature Birth; Ductus Arteriosus, Patent; Sepsis; Asphyxia; Stroke; Hypertension, Pulmonary; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Feasibility study - Healthy neonates: Neonates born with gestational week < 32 weeks, gestational week 32-37 and at term. Will will include 20-30 of each sex in each group.
  Interventions: Device: NeoDoppler - CE certified
- Patients with patent ductus arteriosus (premature infants): Preterm neonates with patent ductus arteriosus (n=20)
  Interventions: Device: NeoDoppler - CE certified
- Different groups of sick neonates: Neonates with different medical conditions such as perinatal asphyxia, stroke, pulmonary hypertension and congenital heart disease will be conducted. We will include 5-30 neonates in each group.
  Interventions: Device: NeoDoppler - CE certified
- Neonates/infants undergoing procedures: Neonates/infants undergoing procedures such as intubation, anesthesia, spinal puncture, peripheral and central arterial and venous catheter. We will include 20-30 neonates.
  Interventions: Device: NeoDoppler - CE certified
- Neonates with infection/sepsis: Infants with infection/sepsis and/or meningitis (n=40).
  Interventions: Device: NeoDoppler - CE certified

INTERVENTIONS:
Device: NeoDoppler - CE certified — The NeoDoppler is small and light weighed constructed as a single element transducer, that can be gently fixed over the fontanelle. The system is fully compatible for cooccurring use with other intensive care equipment for neonates as well as caregiving from the parents. It is capable of measuring cerebral blood flow at different depths of the brain simultaneously. The Doppler velocity measurements arise from a cylindrical volume of tissue. It is therefore less sensitive to the exact position and angle of the probe over the fontanel to target the vessels of interest than standard hand-held Doppler. This means that the NeoDoppler system may be placed by healthcare professionals who do not have specialized training performing diagnostic ultrasound exams of the cerebral vasculature in neonates.

SUMMARY:
Non-invasive tools for monitoring of course of disease are important and necessary in the treatment of pre-term/premature infants and sick neonates. For many years, the ultrasound group in Trondheim has been at the forefront in the development of new ultrasound technology for the diagnosis and monitoring of disease. Several methods previously developed in this research group are today widely used in hospitals around the world. In this project the investigators aim to test a new ultrasound technology that allows continuous monitoring of cerebral blood flow in sick neonates and pre-term children. This technology was CE-certified in October 2022, and in this project the investigators will test the CE-certified version with the newest available approved software.

DETAILED DESCRIPTION:
A new ultrasound technology called NeoDoppler has been developed, which can measure blood flow in the brain over time. The product is approved for clinical use (CE approved). A pilot study, with with inclusion of different patient groups in need of continuous monitoring, will be conducted to map variability of cerebral hemodynamics. These studies include:

1. A feasibility study on healthy preterm- and term born neonates to map what is normal cerebral blood flow in neonates born before gestational week 32, in gestational week 32-37 and at term.
2. A study including preterm neonates with patent ductus arteriosus to look at the connection between the heart's function and the brain's blood flow.
3. Studies of sick neonates including conditions such as perinatal asphyxia, stroke, pulmonary hypertension and congenital heart disease to study how different medical conditions influences cerebral blood flow.
4. A study on cerebral blood flow during ongoing procedures such as intubation, anesthesia, spinal puncture and peripheral and central arterial- and venous catheter.
5. A study of how infection, sepsis and meningitis affects cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Open fontanelle
* Healthy preterm or term born neonates
* Neonates with a medical condition of interest according to the different cohort studies: patent ductus arteriosus, perinatal asphyxia, stroke, pulmonary hypertension, congenital heart condition or infection/sepsis/meningitis
* Neonates in need of procedures

Exclusion Criteria:

* Caregivers not understanding/speaking Norwegian or English
* Caregivers not giving their consent

Ages: 0 Minutes to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates/infants born prematurely or at term that are healthy or that have a medical contentions or that are in need of procedures that are admitted to the maternal ward or neonatal intensive care at St. Olavs Hospital in Trondheim, Norway.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral Doppler velocities (cm/second) | 2 hours - 7 days
  Cerebral Doppler velocities measured in cm/sec is generated by tracing of the Doppler spectrum.

SECONDARY OUTCOMES:
Measurement quality | 2 hours - 7 days
  Quality indicator:
  Defined as a scale from 0-100% where 100% is the best possible Doppler spectrum quality. Values below 80% is below the threshold of good enough quality to be used as valid measurements in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Siri Ann Nyrnes, MD, PhD, Principal Investigator — Childrens Clinic, St. Olavs University Hospital and NTNU; Øyvind Rognmo, PhD, Study Director — Norwegian University of Science and Technology, Trondheim, Norway
Locations (1):
- Children's clinic, St. Olavs University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Anonymous ultrasound data can be shared on reasonable request